CLINICAL TRIAL: NCT04917432
Title: Early and Midterm Outcomes of Intravascular Ultrasound (IVUS) Versus Non-IVUS Guidance in Complex Coronary Chronic Total Occlusion (CTO) Revascularization.
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Assiut University (Other)
Responsible Party: Principal Investigator, Khaled Saber Abdelaal Qayed, Assistant lecturer, Assiut University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: Chronic total occlusion
Record Dates: First submitted 2021-05-27; First posted 2021-06-08 (Actual); Last update posted 2021-06-08 (Actual); Status verified 2021-06

CONDITIONS: Chronic Total Occlusion of Coronary Artery
MeSH Terms: interventions — Ultrasonography, Interventional

STUDY DESIGN:
Who Masked: Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- IVUS guided CTO revascularization (Active Comparator): To assess the effects of IVUS usage in CTO revascularization compared to conventional non-IVUS guided CTO-PCI as regard technical success and procedural success, MACE within 6 months.
  Interventions: Procedure: intravascular ultrasound (IVUS)
- Non-IVUS guided CTO revascularization (Active Comparator): To compare this conventional non-IVUS guided CTO-PCI arm with the other IVUS guided arm as regard technical success and procedural success, MACE within 6 months.
  Interventions: Procedure: Conventional CTO PCI (non-IVUS guided)

INTERVENTIONS:
Procedure: intravascular ultrasound (IVUS) — Intravascular imaging using a specialized catheter delivered through intra-arterial approach to reach the coronaries to guide CTO-PCI procedure and optimize the results after wire crossing.
  Arms: IVUS guided CTO revascularization
Procedure: Conventional CTO PCI (non-IVUS guided) — Non-IVUS guided CTO PCI for wiring but may be used for results optimization after wire crossing
  Arms: Non-IVUS guided CTO revascularization

SUMMARY:
Various CTO percutaneous coronary intervention (PCI) studies defined CTO as as a substantial atherosclerotic blockage with >3 months duration of TIMI (Thrombolysis in Myocardial Infarction) 0 flow other than via collaterals. Following CTO-PCI, various well-established therapeutic benefits have been extensively acknowledged, such as improved angina frequency score and quality of life score from the Seattle Angina Questionnaire (SAQ). Patients are currently referred for CTO PCI to relieve symptoms, reduce ischemia load, or pursue full revascularization to improve left ventricular ejection fraction (LVEF) CTO-PCI is one of the most difficult procedures in interventional cardiology today. Although IVUS has been demonstrated to improve long-term results during CTO PCI when used for stent optimization, its impact on crossing has received little research. IVUS imaging can aid in the resolution of proximal cap ambiguity by determining the position of the main branch and determining the position of the guidewire during CTO crossing efforts both antegrade and retrograde. For the reverse controlled antegrade and retrograde tracking and dissection (reverse CART) procedure, IVUS can help establish the best balloon size. In addition, imaging guidance can help in balloon and stent sizing, as well as stent expansion and strut apposition.

The function of IVUS in CTO PCI has been a source of contention among the four major CTO schools hybrid algorithms. The importance of IVUS-guided entry in overcoming proximal cap uncertainty was underlined in the Asia Pacific algorithm. Furthermore, IVUS-guided wiring, limited subintimal tracking and re-entry are incorporated in the algorithm as alternatives, but only as last resorts. After performing dual coronary injections, the North American hybrid method evaluates four angiographic characteristics, the first of which is a clear understanding of the proximal cap placement utilising angiography or IVUS. They also explain how IVUS guidance can help with reverse CART by allowing for the proper balloon size selection. When proximal cap ambiguity is found in the Euro CTO club algorithm, antegrade procedures such as IVUS-guided puncture and scratch and go technique are performed. When using a primary retrograde approach, the probability of antegrade passing with IVUS guidance and parallel wiring, as well as the advantage of a shorter guide wire crossing time when employing an antegrade route alone, must be incorporated in the Japanese algorithm.

ELIGIBILITY:
Inclusion Criteria:

- All coronary CTO patients in whom coronary anatomy is defined by coronary CT and/or Coronary angiography provided that:- CTO defined as heavy atherosclerotic occlusion with TIMI (Thrombolysis in Myocardial Infarction) 0 flow other than via collaterals for >3 months and they are symptomatic despite optimal medical therapy and/or positive high risk stress modality.

Exclusion Criteria:

* Acute coronary syndrome within 3 months.
* Patients with renal insufficiency (eGFR < 60 ml/kg/m2, serum creatinine ≥ 2.5 mg/dL, or on regular dialysis).
* Patients with expected post CTO-PCI procedure SYNTAX >10.
* Hemodynamically unstable patients.

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 70 (Estimated)
Dates: Start 2022-09-01 (Estimated); Primary Completion 2024-09-30 (Estimated); Study Completion 2025-09-30 (Estimated)

PRIMARY OUTCOMES:
Technical success | Within three to six hours
  Restoration of antegrade flow with residual stenosis below 30% assessed using IVUS by measuring the minimal lumenal area in mm2
procedural success | within three days
  technical success without in-hospital MACE (death, myocardial infarction, need for urgent PCI or CABG and stroke).
major adverse cardiovascular events (MACE) | within six months
  death, myocardial infarction, repeat target vessel revascularization with either PCI or coronary artery bypass graft surgery and stroke

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Galassi AR, Werner GS, Boukhris M, Azzalini L, Mashayekhi K, Carlino M, Avran A, Konstantinidis NV, Grancini L, Bryniarski L, Garbo R, Bozinovic N, Gershlick AH, Rathore S, Di Mario C, Louvard Y, Reifart N, Sianos G. Percutaneous recanalisation of chronic total occlusions: 2019 consensus document from the EuroCTO Club. EuroIntervention. 2019 Jun 20;15(2):198-208. doi: 10.4244/EIJ-D-18-00826. PMID 30636678
- [Background] Hong SJ, Kim BK, Shin DH, Kim JS, Hong MK, Gwon HC, Kim HS, Yu CW, Park HS, Chae IH, Rha SW, Lee SH, Kim MH, Hur SH, Jang Y; K-CTO Registry. Usefulness of intravascular ultrasound guidance in percutaneous coronary intervention with second-generation drug-eluting stents for chronic total occlusions (from the Multicenter Korean-Chronic Total Occlusion Registry). Am J Cardiol. 2014 Aug 15;114(4):534-40. doi: 10.1016/j.amjcard.2014.05.027. Epub 2014 Jun 6. PMID 25001153
- [Background] Park Y, Park HS, Jang GL, Lee DY, Lee H, Lee JH, Kang HJ, Yang DH, Cho Y, Chae SC, Jun JE, Park WH. Intravascular ultrasound guided recanalization of stumpless chronic total occlusion. Int J Cardiol. 2011 Apr 14;148(2):174-8. doi: 10.1016/j.ijcard.2009.10.052. Epub 2009 Nov 26. PMID 19942305
- [Background] Dai J, Katoh O, Kyo E, Tsuji T, Watanabe S, Ohya H. Approach for chronic total occlusion with intravascular ultrasound-guided reverse controlled antegrade and retrograde tracking technique: single center experience. J Interv Cardiol. 2013 Oct;26(5):434-43. doi: 10.1111/joic.12066. PMID 24106742
- [Background] Estevez-Loureiro R, Ghione M, Kilickesmez K, Agudo P, Lindsay A, Di Mario C. The role for adjunctive image in pre-procedural assessment and peri-procedural management in chronic total occlusion recanalisation. Curr Cardiol Rev. 2014 May;10(2):120-6. doi: 10.2174/1573403x10666140331143731. PMID 24694101
- [Background] Kalogeropoulos AS, Alsanjari O, Davies JR, Keeble TR, Tang KH, Konstantinou K, Vardas P, Werner GS, Kelly PA, Karamasis GV. Impact of Intravascular Ultrasound on Chronic Total Occlusion Percutaneous Revascularization. Cardiovasc Revasc Med. 2021 Dec;33:32-40. doi: 10.1016/j.carrev.2021.01.008. Epub 2021 Jan 12. PMID 33461936